CLINICAL TRIAL: NCT06275048
Title: The Effects of Oral Contraceptive Use on Grip Strength and Neuromuscular Activation During Short-Term Immobilization of the Wrist/Hand
Brief Title: The Influence of Oral Contraceptives During Disuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Matt Stock, Associate Professor, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006302
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Oral Contraceptives; Rehabilitation; Menstrual Cycle; Physical Therapy
Keywords: oral contraceptives; menstrual cycle; immobilization; weakness; rehabilitation
MeSH Terms: conditions — Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wrist/hand immobilization (Experimental): Participants will have their wrist and hand immobilized using a rigid splint continuously for 7 days. The splint will restrict all wrist and hand movement and must be worn at all times for the full 7 day period, and may only be removed under supervision of the research participants.
  Interventions: Other: Wrist/hand immobilization

INTERVENTIONS:
Other: Wrist/hand immobilization — Study participants will have their left wrist/hand immobilized with a splint for 7 days. The splint will be worn 24 hours per day.

SUMMARY:
Studies across various sports and physical activities have consistently shown that females incur more injuries compared to their male counterparts, but the underlying reasons for this disparity remain poorly understood. While differences in hormone levels between males and females have been speculated to play a role, very little rigorous research has been conducted to directly examine potential connections between sex hormones and injury risk. Specifically, females have been shown to be at greater risk for hand and wrist injuries. The higher injury incidence begins at puberty and persists across the lifespan, suggesting a link to hormonal factors. However, significant gaps remain in understanding the relationships between the menstrual cycle, exogenous hormones from birth control, and risk factors for sports-related injury in females. The purpose of this study is to examine changes in muscle strength and neuromuscular activation among females using monophasic oral contraceptives, females not using oral contraceptives, and males during one week of wrist/hand immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Right handed males and females
* Ages 18-35 years
* For females, consistent use of monophasic oral contraceptives for the previous 6 months OR having completely refrained from contraceptives for the previous 6 months.

Exclusion Criteria:

* Gender identity inconsistent with biological sex (due to the influence that drugs used for gender reassignment may have)
* Females that are amenorrheic (lack of menstruation for ≥3 consecutive cycles) or oligomenorrheic (menstrual cycle length ≤36 days)
* Menstrual cycle irregularities among females not using oral contraceptives (regularity defined as every 21 to 35 days and/or at least 5 periods in the last six months)
* Any contraceptive use other than monophasic oral contraceptives within the last 6 months
* Monophasic oral contraceptives that has been inconsistent over the previous 6 months
* Score of greater than 2/5 on question 9, or a score of greater than 1/5 on question 10 or 11 on the quick Disabilities of the Arm, Shoulder and Hand outcome measure indicating pain/discomfort of the upper extremities (shoulder, elbow, wrist, hand)
* Dominant hand is the left hand
* Body Mass Index less than 18.5 kg/m2 or greater than 29.9 kg/m2
* Current depression or anxiety
* History of musculoskeletal injury, pain, or surgery of the elbow, wrist, or hand
* Unwillingness to avoid upper-body exercise during Phase 1
* Unwillingness to avoid exercise and alcohol 24 hours prior to each testing visit.
* Neuromuscular disease (e.g., Multiple Sclerosis, amyotrophic lateral sclerosis, Parkinson's)
* Metabolic disease (e.g., diabetes, thyroid disorder, metabolic syndrome)
* Personal or family history of blood clots
* Trouble using or controlling muscles
* History of cancer
* History of stroke
* History of heart attack
* History of arthritis
* Allergy to rubbing alcohol
* Lack of transportation to and from the laboratory
* Current or planned pregnancy (within the next three months)
* Implant of any kind
* The use of medications that may increase the risk of blood clots (i.e., corticosteroids such as prednisone, testosterone and anabolic steroids, selective estrogen receptor modulators like tamoxifen, aromatase inhibitors including anastrozole, thalidomide and lenalidomide, erythropoiesis-stimulating agents such as epoetin alfa, antipsychotics like chlorpromazine, antidepressants including paroxetine, various cancer chemotherapies, immune modulating drugs, antivirals such as ritonavir, and tamoxifen).
* The use of creatine monohydrate and beta alanine supplementation within the previous 6 months.
* The use of any medication or supplement that could influence hormone levels within the previous 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males and females. Gender identity must be consistent with biological sex.
Enrollment: 41 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Grip Strength | Grip strength will be tested weekly for at least 3 weeks (i.e., baseline, post-immobilization, post 1 week recovery). Testing will continue every week following immobilization until grip strength has returned to baseline levels.
  Maximal force (N) will be measured during a grip strength test

SECONDARY OUTCOMES:
Muscle activation | Grip strength will be tested weekly for at least 3 weeks (i.e., baseline, post-immobilization, post 1 week recovery). Testing will continue every week following immobilization until grip strength has returned to baseline levels.
  Surface electromyographic amplitude of hand and wrist muscles will be measured during the maximal grip tests.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make de-identified individual participant data (IPD) from this study available to other researchers once the primary analysis is completed and the study results have been published. The data will be shared in a manner that protects participant confidentiality and adheres to applicable laws and regulations.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available beginning 1 year after the study completion date.
Access Criteria: Researchers must submit a methodologically sound proposal outlining their planned analysis of the data. Proposals will be reviewed and approved by an independent panel appointed by the Principal Investigator. Requests should be sent to matt.stock@ucf.edu